CLINICAL TRIAL: NCT04916769
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 3-PERIOD, 6-SEQUENCE, CROSSOVER STUDY TO EVALUATE THE BIOAVAILABILITY OF BOSUTINIB ADMINISTERED AS CAPSULE CONTENTS MIXED WITH APPLESAUCE OR YOGURT RELATIVE TO INTACT CAPSULES IN HEALTHY PARTICIPANTS UNDER FED CONDITION
Brief Title: Bioavailability of Bosutinib Administered as Capsule Contents Mixed With Applesauce or Yogurt Relative to Intact Capsules Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1871063; 2021-000500-38 (EudraCT Number)
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: Bioavailability; bosutinib; Maximum Observed Plasma Concentration (Cmax); Area Under the Curve (AUC)
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Intervention Model Description: A Phase 1, open-label, randomized, single dose, 3-period, 6-sequence, crossover study in healthy participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bosutinib capsule contents mixed with applesauce (Experimental): Bosutinib capsule contents mixed with applesauce to healthy participants
  Interventions: Drug: Bosutinib capsule
- Bosutinib capsule contents mixed with yogurt (Experimental): Bosutinib capsule contents mixed with yogurt to healthy participants
  Interventions: Drug: Bosutinib capsule
- Bosutinib intact capsules (Active Comparator): Bosutinib intact capsules to healthy participants
  Interventions: Drug: Bosutinib capsule

INTERVENTIONS:
Drug: Bosutinib capsule — 500 mg dose of bosutinib capsule contents mixed with applesauce
  Arms: Bosutinib capsule contents mixed with applesauce
Drug: Bosutinib capsule — 500 mg dose of bosutinib capsule contents mixed with yogurt
  Arms: Bosutinib capsule contents mixed with yogurt
Drug: Bosutinib capsule — 500 mg dose of intact bosutinib capsules
  Arms: Bosutinib intact capsules

SUMMARY:
This study is intended to estimate the relative bioavailability of a single 500 mg dose of bosutinib when administered as capsule contents mixed with applesauce or yogurt to intact capsules under fed condition in adult healthy participants. The comparisons will be performed using the pharmacokinetic parameters that define the rate and extent of absorption, those are Cmax and AUC. Statistical analyses will be performed comparing these parameters calculated after administration of a single 500 mg dose with the intact capsule formulation (100 mg x 5) as the Reference treatment and the capsule contents mixed with applesauce or yogurt (100 mg x 5) as the Test treatments.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non childbearing potential and/or male participants must be 18 to 54 years of age, inclusive, at the time of signing the informed consent document (ICD).
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease.
* Any condition possibly affecting drug absorption.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

  1. estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) < 90 mL/min/1.73 m2;
  2. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > upper limit of normal (ULN);
  3. Serum (total and direct) bilirubin level > ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN;
  4. Amylase and lipase levels > ULN.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1871063

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants were assigned to the study intervention, 16 of whom received all the 3 randomized treatment by sequence and completed the study.
Groups:
- Sequence 1: Treatment C=>Treatment A =>Treatment B; Sequence 2: Treatment B=>Treatment C =>Treatment A; Sequence 3: Treatment A=>Treatment B =>Treatment C; Sequence 4: Treatment B=>Treatment A =>Treatment C; Sequence 5: Treatment A=>Treatment C =>Treatment B; Sequence 6: Treatment C=>Treatment B =>Treatment A: Treatment A: Bosutinib 500 mg single dose was administered as capsule contents mixed with 45 mL applesauce. Treatment B: Bosutinib 500 mg single dose was administered as capsule contents mixed with 45 mL yogurt. Treatment C: Bosutinib 500 mg single dose was administered as intact capsules. There were at least 14 days between successive bosutinib doses.
Period: Period 1
Arm/Group | Sequence 1: Treatment C=>Treatment A =>Treatment B | Sequence 2: Treatment B=>Treatment C =>Treatment A | Sequence 3: Treatment A=>Treatment B =>Treatment C | Sequence 4: Treatment B=>Treatment A =>Treatment C | Sequence 5: Treatment A=>Treatment C =>Treatment B | Sequence 6: Treatment C=>Treatment B =>Treatment A
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sequence 1: Treatment C=>Treatment A =>Treatment B | Sequence 2: Treatment B=>Treatment C =>Treatment A | Sequence 3: Treatment A=>Treatment B =>Treatment C | Sequence 4: Treatment B=>Treatment A =>Treatment C | Sequence 5: Treatment A=>Treatment C =>Treatment B | Sequence 6: Treatment C=>Treatment B =>Treatment A
Started | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 2 | 3 | 3 | 3 | 2
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: Treatment C=>Treatment A =>Treatment B | Sequence 2: Treatment B=>Treatment C =>Treatment A | Sequence 3: Treatment A=>Treatment B =>Treatment C | Sequence 4: Treatment B=>Treatment A =>Treatment C | Sequence 5: Treatment A=>Treatment C =>Treatment B | Sequence 6: Treatment C=>Treatment B =>Treatment A
Started | 3 | 2 | 3 | 3 | 3 | 2
Completed | 3 | 2 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention.
Groups:
- Entire Study Population: Includes all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 32.0 [21 to 54]
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 3
  26-35 years | 8
  36-45 years | 5
  Older than 45 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — For the "sex" category, the participant count for one of the genders was very low, which if reported would risk re-identification of the participant. Hence, data was not reported for this baseline characteristics.
  Male | NA — For the "sex" category, the participant count for one of the genders was very low, which if reported would risk re-identification of the participant. Hence, data was not reported for this baseline characteristics.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for Bosutinib
Description: AUCinf was calculated as [AUClast+(Clast*/kel)], where AUClast is the area under the plasma concentration-time profile from time 0 to the time of the Clast, Clast is the last quantifiable concentration, Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: Total number of participants received treatment and had bosutinib pharmacokinetic (PK) parameter contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram•hour per milliliter (ng•hr/mL)
Groups:
- Bosutinib 500 mg Capsule Contents + Applesauce 45 mL: Bosutinib 500 mg single dose was administered as capsule contents mixed with 45 mL applesauce.
- Bosutinib 500 mg Capsule Contents + Yogurt 45 mL: Bosutinib 500 mg single dose was administered as capsule contents mixed with 45 mL yogurt.
- Bosutinib 500 mg Intact Capsule: Bosutinib 500 mg single dose was administered as intact capsules.
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 17
nanogram•hour per milliliter (ng•hr/mL) | 3312 (28) | 3205 (23) | 3161 (32)
Statistical Analysis 1: Comparison: Bosutinib 500 mg Capsule Contents + Applesauce 45 mL vs Bosutinib 500 mg Intact Capsule; Natural logarithm-transformed bosutinib AUCinf was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Bosutinib 500 mg capsule contents + applesauce 45 mL [Test] - Bosutinib 500 mg intact capsule [Reference]) and corresponding 90% confidence intervals (CIs) were obtained from the model; Test type: Equivalence — The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. The ratio of adjusted geometric means and 90% confidence interval were expressed as percentages; ratio of ajusted geometric means = 106.27, 90% CI 2-sided [97.76 to 115.53]
Statistical Analysis 2: Comparison: Bosutinib 500 mg Capsule Contents + Yogurt 45 mL vs Bosutinib 500 mg Intact Capsule; Natural logarithm-transformed bosutinib AUCinf was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Bosutinib 500 mg capsule contents + yogurt 45 mL [Test] - Bosutinib 500 mg intact capsule [Reference]) and corresponding 90% CIs were obtained from the model; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ratio of adjusted geometric means = 101.93, 90% CI 2-sided [93.97 to 110.56]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Bosutinib
Description: Cmax was the maximum observed plasma concentration. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: Total number of participants received treatment and had bosutinib PK parameter contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 17
nanogram per milliliter (ng/mL) | 126.5 (31) | 126.1 (27) | 132.0 (33)
Statistical Analysis 1: Comparison: Bosutinib 500 mg Capsule Contents + Applesauce 45 mL vs Bosutinib 500 mg Intact Capsule; Natural logarithm-transformed bosutinib Cmax was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Bosutinib 500 mg capsule contents + applesauce 45 mL [Test] - Bosutinib 500 mg intact capsule [Reference]) and corresponding 90% CIs were obtained from the model; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ratio of adjusted geometric means = 96.82, 90% CI 2-sided [86.37 to 108.53]
Statistical Analysis 2: Comparison: Bosutinib 500 mg Capsule Contents + Yogurt 45 mL vs Bosutinib 500 mg Intact Capsule; Natural logarithm-transformed bosutinib Cmax was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Bosutinib 500 mg capsule contents + yogurt 45 mL [Test] - Bosutinib 500 mg intact capsule [Reference]) and corresponding 90% CIs were obtained from the model; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ratio of adjusted geometric means = 95.39, 90% CI 2-sided [85.34 to 106.61]

3. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for Bosutinib
Description: AUClast was the area under the concentration-time curve from time 0 to the time of the last quantifiable concentration. Linear/Log trapezoidal method was used to determine AUClast. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: Total number of participants received treatment and had bosutinib PK parameter contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram•hour per milliliter (ng•hr/mL)
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 17
nanogram•hour per milliliter (ng•hr/mL) | 3150 (28) | 3055 (23) | 3009 (33)
Statistical Analysis 1: Comparison: Bosutinib 500 mg Capsule Contents + Applesauce 45 mL vs Bosutinib 500 mg Intact Capsule; Natural logarithm-transformed bosutinib AUClast was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Bosutinib 500 mg capsule contents + applesauce 45 mL [Test] - Bosutinib 500 mg intact capsule [Reference]) and corresponding 90% CIs were obtained from the model; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ratio of adjusted geometric means = 106.23, 90% CI 2-sided [97.54 to 115.68]
Statistical Analysis 2: Comparison: Bosutinib 500 mg Capsule Contents + Yogurt 45 mL vs Bosutinib 500 mg Intact Capsule; Natural logarithm-transformed bosutinib AUClast was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Bosutinib 500 mg capsule contents + yogurt 45 mL [Test] - Bosutinib 500 mg intact capsule [Reference]) and corresponding 90% CIs were obtained from the model; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ratio of adjusted geometric means = 102.08, 90% CI 2-sided [93.95 to 110.91]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Bosutinib
Description: Tmax was the time to reach maximum observed plasma concentration and was observed directly from data as time of the first occurrence.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: Total number of participants received treatment and had bosutinib PK parameter contributing to the summary statistics.
Measure: Median (Full Range); unit: hour
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 17
hour | 6.00 [2.00 to 8.02] | 6.00 [2.00 to 8.00] | 6.00 [3.00 to 12.0]

5. Secondary Outcome: Apparent Clearance After Oral Dose (CL/F) for Bosutinib
Description: CL/F was the apparent clearance after oral dose and was determined as dose/AUCinf. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: Total number of participants received treatment and had bosutinib PK parameter contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 17
liter/hour | 151.0 (28) | 156.0 (23) | 158.1 (32)

6. Secondary Outcome: Apparent Volume of Distribution After Oral Dose (Vz/F) for Bosutinib
Description: Vz/F was the apparent volume of distribution after oral dose. It was determined as dose/(AUCinf × kel), where kel was the terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration time curve. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: Total number of participants received treatment and had bosutinib PK parameter contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 17
liter | 7903 (31) | 8106 (28) | 8145 (41)

7. Secondary Outcome: Terminal Phase Half-life (t½ ) for Bosutinib
Description: t½ was the terminal elimination plasma half-life. It was determined as Loge(2)/kel, where kel was the terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: Total number of participants received treatment and had bosutinib PK parameter contributing to the summary statistics.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 17
hour | 36.46 (3.7067) | 36.30 (4.6893) | 36.02 (4.9889)

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory tests included hematology tests, chemistry tests, and urinalysis tests.
Time Frame: Post first dose and up to Day 7 in Period 3, or at early termination/discontinuation.
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 18
Participants | 8 | 11 | 11

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Severe Adverse Events (AEs), and Serious Adverse Events (SAEs)
Description: TEAEs are those with initial onset or that worsen in severity after the first dose of the study medication. All AEs in the table below were TEAEs. An SAE is any untoward medical occurrence at any dose that: results in death; is life threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect; or that is considered to be an important medical event. Severe AEs were defined as AEs that interfered significantly with participant's usual function. Both SAEs and severe AEs were according to the investigator's assessment.
Time Frame: Up to 12 weeks
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
Number analyzed (Participants) | 16 | 17 | 18
Participants
  Participants with TEAEs | 11 | 14 | 15
  Participants with SAEs | 0 | 0 | 0
  Participants with severe AEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The analysis of adverse events included all participants who received at least 1 dose of the randomized study treatment.
Arm/Group | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL | Bosutinib 500 mg Intact Capsule
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 11/16 | 14/17 | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 500 mg Capsule Contents + Applesauce 45 mL (N=16) | Bosutinib 500 mg Capsule Contents + Yogurt 45 mL (N=17) | Bosutinib 500 mg Intact Capsule (N=18)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 11 | 10
Eructation (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 6 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 3 | 3 | 2
Feeling of body temperature change (General disorders) | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 2 | 0
Vessel puncture site reaction (General disorders) | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT04916769/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04916769/SAP_001.pdf